CLINICAL TRIAL: NCT02354131
Title: Part 1: AVANOVA1 - A Phase I Study to Evaluate the Safety and Tolerability of Bevacizumab-niraparib Combination Therapy and Determine the Recommended Phase 2 Dose (RP2D) in Women With Platinum-sensitive Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer Part 2: AVANOVA2 - A Two-arm, Open-label, Phase II Randomized Study to Evaluate the Efficacy of Niraparib Versus Niraparib-bevacizumab Combination in Women With Platinum-sensitive Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer.
Brief Title: Niraparib Versus Niraparib-bevacizumab Combination in Women With Platinum-sensitive Epithelial Ovarian Cancer
Acronym: AVANOVA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Gynecologic Cancer Intergroup (GCIG) (Other); University of Utah (Other); Massachusetts General Hospital (Other); Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-OV24-NSGO/AVANOVA
Record Dates: First submitted 2015-01-25; First posted 2015-02-03 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Niraparib; Bevacizumab; PARP; Phase 2 randomized
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Niraparib monotherapy (Experimental): Niraparib mono therapy until progression
  Interventions: Drug: Niraparib
- Niraparib-bevacizumab combination (Experimental): Niraparib-bevacizumab combination therapy until progression
  Interventions: Drug: Niraparib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Niraparib — Niraparib versus Bevacizumab-Niraparib combo
Drug: Bevacizumab
  Arms: Niraparib-bevacizumab combination

SUMMARY:
Part 1 (Phase 1): safety and tolerability of bevacizumab-Niraparib combination Part 2 (Randomized Phase 2): to compare Progression-Free Survival (PFS)

PARP inhibitors are active as monotherapy to treat patients with recurrent ovarian cancer; the strongest activity being observed in the platinum sensitive, gBRCAmut subgroup as well as in gBRCAwt, HRD population but also in HRD negative disease.

In the same population there is level one evidence that bevacizumab is beneficial. And a phase two randomized study has indicated that combination of a PARP inhibitor with anti-angiogenic drug is superior to PARP inhibitor alone.

The question is:

Is niraparib combined with bevacizumab superior to niraparib? The comparison of tolerability and efficacy of niraparib-bevacizumab combination against niraparib.

DETAILED DESCRIPTION:
Part 1: This is a single-centre, phase 1a, open-label, dose-escalation study to evaluate the safety and tolerability of bevacizumab-niraparib combination and determine the RP2D in patients with platinum-sensitive epithelial ovarian, fallopian tube, or primary peritoneal cancer.

The standard 3+3 design will be used. Part 2: (n=94) This multicenter, prospective, open-label, randomized phase 2 study is evaluating the efficacy of niraparib against niraparib-bevacizumab combination in Women with platinum-sensitive epithelial ovarian, fallopian tube, or primary peritoneal cancer.

Stratification: Patients are stratified according to:

1. HRD status (positive/negative)
2. Treatment-Free interval to prior therapy (6-12 months > 12 months) Randomization: 1:1 randomization

Study arms: Patients are randomized to one of the two treatment arms:

Arm 1: Niraparib monotherapy until progression. Arm 2: Niraparib-bevacizumab combination therapy until progression.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion only if all of the following criteria are fulfilled:

1. Recurrent platinum-sensitive epithelial ovarian, fallopian tube, or peritoneal cancer (platinum sensitivity defined as no recurrence within 6 months of last receipt of platinum/chemotherapy).
2. High-grade serious or high-grade endometrioid histology.
3. Patient consents to perform HRD test.

   * Patients with known BRCA status: BRCA positive patients must submit the tissue for HRD test, though these patients need not to wait for HRD test results and can be randomized in HRD positive stratum.
   * If tumor tissue is not sufficient to perform HRD test: these patients shall be randomized in HRD negative stratum as HRD unknown.
4. Prior line of therapy: Patients must have received platinum-containing therapy for primary disease.

   * No limits on number of platinum-based therapies. Population of patients who has previously received ≥ 3 lines of therapy for relapsed disease will be capped at 40%.
   * Up to one non-platinum-based line of therapy in recurrent setting.
   * Patients who are treated with bevacizumab just prior to entering in the trial must not have progressed under or within 3 months after bevacizumab.
   * Patients may have participated in a PARP inhibitor trial as first-line maintenance therapy and have not progressed within 3 months after PARP/placebo. Patients who received PARP inhibitor after relapse (definitive or maintenance therapy) are not eligible.
5. Target group: Age 18+
6. Histological confirmed ovarian, fallopian tube or peritoneal cancers
7. Patients must give informed consent
8. Patients may have undergone primary or interval debulking surgery
9. Patients may have received bevacizumab though no other prior use of anti-angiogenic therapy
10. Patients may have received a PARP inhibitor as first-line maintenance therapy.
11. Patients must have disease that is measurable according to RECIST or assessable according to the GCIG criteria
12. The patient agrees to complete PROs (QoL questionnaire) during study treatment AND at one additional time point 8 weeks following progression of disease
13. ECOG performance status 0-2
14. Adequate organ function

    * Absolute neutrophil count (ANC) ≥1,5 x 109/L
    * Platelets >100 x 109/L
    * Hemoglobin ≥ 9g/dl
    * Serum creatinine ≤1.5x upper limit of normal (ULN) or calculated creatinine clearance ≥50mL/min using Cockcroft-Gault formula
    * Total bilirubin ≤1.5x ULN
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5x ULN unless liver metastases are present, in which case they must be ≤5x ULN.
15. Able to take oral medications
16. Life expectancy of at least 12 weeks
17. Patients must fulfill all inclusions criteria and according to investigator fit to receive niraparib and/or bevacizumab.
18. Women of childbearing potential must use adequate birth control for the duration of study participation

Exclusion Criteria:

A patient will not be eligible for inclusion if any of the following criteria are fulfilled:

1. Ovarian sarcomas, small cell carcinoma with neuroendocrine differentiation, non-epithelial cancers and cancer types not mentioned in the inclusion criteria
2. Concurrent cancer therapy
3. Concurrent treatment with an investigational agent or participation in another clinical trial
4. Major injuries or surgery within the past 21 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period
5. Previous malignant disease: patients are not eligible for the study if diagnosis, detection or treatment of invasive cancer (other than ovarian cancer; with the exception of basal or squamous cell carcinoma of the skin that was definitively treated) was detected within 2 years prior to randomization
6. Active infections or other serious underlying significant medical illness, abnormal laboratory finding or psychiatric illness/social situation that would, in the Investigator's judgment, makes the patient inappropriate for this study
7. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
8. History of bowel obstruction, including sub-occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess. Evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction
9. Known contraindications to PARP inhibitors or VEGF directed therapy
10. Known uncontrolled hypersensitivity to the investigational drugs
11. History of major thromboembolic event defined as:

    * Uncontrolled pulmonary embolism (PE)
    * Deep venous thrombosis (DVT)
    * Other related conditions, though patients with stable therapeutic anticoagulation for more than three months prior randomization are eligible for this study. This also apply to PE & DVT.
12. History of a cerebral vascular accident, transient ischemic attack or subarachnoid hemorrhage within the past 3 months
13. History of clinically significant hemorrhage in the past 3 months
14. Uncontrolled and/or symptomatic CNS metastasis or leptomeningeal carcinomatosis (Dexamethasone/prednisone therapy will be allowed if administered as stable dose for at least one month prior randomization)
15. Significant cardiovascular diseases, including uncontrolled hypertension, clinically relevant cardiac arrhythmia, unstable angina or myocardial infarction within 6 months prior to randomization, congestive heart failure > NYHA III, severe peripheral vascular disease, QT prolongation >470 msec ,clinically significant pericardial effusion
16. Pregnancy or breastfeeding. Patients with preserved reproductive capacity, unwilling to use a medically acceptable method of contraception for the duration of the trial and for 3 months afterwards.
17. Radiographic evidence of cavitation or necrotic tumors with invasion of adjacent major blood vessels
18. Active or chronic hepatitis C and/or B infection
19. Persistence of clinically relevant therapy related toxicity from previous chemotherapy
20. Proteinuria as demonstrated by: (a) urine protein: creatinine (UPC) ratio >/= 1.0 at screening OR (b) urine dipstick for proteinuria >/=2+ (patients discovered to have >/=2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hr urine collection and must demonstrate </=1g of protein in24 hours to be eligible
21. Patients must not have any known history of MDS
22. Patients must not have known persistent (> 4 weeks) ≥ Grade 2 hematological toxicity from prior cancer therapy
23. Patients must not have known ≥ Grade 3 thrombocytopenia or anemia with the last chemotherapy regimen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 30 months
  This is pick the winer trial. The best arm will be used for phase 3 trial against standard of care.

SECONDARY OUTCOMES:
Disease Control Rate | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor R Mirza, MD, Study Chair — Nordic Society of Gynaecological Oncology - Clinical Trials Unit
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Rigshospitalet, Copenhagen, Region Sjælland, Denmark

REFERENCES:
- [Derived] Korsholm LM, Kjeldsen M, Perino L, Mariani L, Nyvang GB, Kristensen E, Bagger FO, Mirza MR, Rossing M. Combining Homologous Recombination-Deficient Testing and Functional RAD51 Analysis Enhances the Prediction of Poly(ADP-Ribose) Polymerase Inhibitor Sensitivity. JCO Precis Oncol. 2024 Feb;8:e2300483. doi: 10.1200/PO.23.00483. PMID 38427930
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Mirza MR, Avall Lundqvist E, Birrer MJ, dePont Christensen R, Nyvang GB, Malander S, Anttila M, Werner TL, Lund B, Lindahl G, Hietanen S, Peen U, Dimoula M, Roed H, Or Knudsen A, Staff S, Krog Vistisen A, Bjorge L, Maenpaa JU; AVANOVA investigators. Niraparib plus bevacizumab versus niraparib alone for platinum-sensitive recurrent ovarian cancer (NSGO-AVANOVA2/ENGOT-ov24): a randomised, phase 2, superiority trial. Lancet Oncol. 2019 Oct;20(10):1409-1419. doi: 10.1016/S1470-2045(19)30515-7. Epub 2019 Aug 29. PMID 31474354
- [Derived] Mirza MR, Bergmann TK, Mau-Sorensen M, Christensen RD, Avall-Lundqvist E, Birrer MJ, Jorgensen M, Roed H, Malander S, Nielsen F, Lassen U, Brosen K, Bjorge L, Maenpaa J. A phase I study of the PARP inhibitor niraparib in combination with bevacizumab in platinum-sensitive epithelial ovarian cancer: NSGO AVANOVA1/ENGOT-OV24. Cancer Chemother Pharmacol. 2019 Oct;84(4):791-798. doi: 10.1007/s00280-019-03917-z. Epub 2019 Aug 2. PMID 31375879